CLINICAL TRIAL: NCT05511675
Title: The Effect of Cold Application on the Hemostasis, Extremity Pain And Terumo Band Usage After Transradial Angiography
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duzce University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: DuzceU-ismail-01
Record Dates: First submitted 2022-08-18; First posted 2022-08-23 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Radial Artery; Pain; Local Application / Packing Too Cold; Hemostasis; Angiography
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (No Intervention): Patients who are in the control group will receive standard clinical care and pain level and hematoma condition will be recorded. In addition usage time of the TR band will be in accordance with the manufacturer's guidelines and will be recorded with the help of a chronometer.
- experimental group I (Experimental): Study group I patients will have cold application twice for a twenty minute period each time. For study group I extremity pain and hematoma will be followed and the TR band will be removed after one and a half hours.
  Interventions: Device: cold application
- experimental group II (Experimental): Study group II patients will have cold application twice for a twenty minute period each time and extremity pain and hematoma will be followed but the TR band will be removed in accordance with manufacturer's guidelines as in the control group.
  Interventions: Device: cold application

INTERVENTIONS:
Device: cold application — ISO-BALL
  Arms: experimental group I; experimental group II

SUMMARY:
According to the World Health Organization data, approximately 17.9 million people die every year due to heart disease. 85% of these deaths are due to heart attack and blocked blood vessels. The Turkish Statistical Institute reports that circulatory system diseases took the first place among the causes of death with 38.4%, while ischemic heart diseases constituted 39.7% of these deaths in 2018. Transradial angiography is used for the purpose of scanning and treatment of coronary arteries both in Turkey and in other countries of the world.

Aim: After transradial angiography, Terumo (TR) band is used as a common device which is provides pneumatical hemostasis. This study aims to reduce usage time of the TR band, a decrease of hematoma formation and a reduction in the level of extremities pain experienced as a result of transradial angiography, thanks to using the TR band together with cold application.

DETAILED DESCRIPTION:
According to the World Health Organization data, approximately 17.9 million people die every year due to heart disease. 85% of these deaths are due to heart attack and blocked blood vessels. The Turkish Statistical Institute reports that circulatory system diseases took the first place among the causes of death with 38.4%, while ischemic heart diseases constituted 39.7% of these deaths in 2018. Transradial angiography is used for the purpose of scanning and treatment of coronary arteries both in Turkey and in other countries of the world.

Aim: After transradial angiography, Terumo (TR) band is used as a common device which is provides pneumatical hemostasis. This study aims to reduce usage time of the TR band, a decrease of hematoma formation and a reduction in the level of extremities pain experienced as a result of transradial angiography, thanks to using the TR band together with cold application.

Method: This study is planned to be carried out among the patients who apply for transradial angiography between 15.09.2022 and 15.01.2023 at Düzce University Health Application and Research Center. This study will consist of a control and two experimental groups. This study is planned to be done as a single blind randomised control trial and will use equal samples block randomisation design. The study is planned to comprise of 120 patients, 40 patients in each group, taking into account possible losses. Samples number is to be calculated via G-power 3.1.9.7 programme.

Patients who are in the control group will receive standard clinical care and pain level and hematoma condition will be recorded. In addition usage time of the TR band will be in accordance with the manufacturer's guidelines and will be recorded with the help of a chronometer.

Study group I and group II patients will have cold application twice for a twenty minute period each time. For study group I extremity pain and hematoma will be followed and the TR band will be removed after one and a half hours.

Whereas, for study group II extremity pain and hematoma will be followed but the TR band will be removed in accordance with manufacturer's guidelines as in the control group.

Data accumulation methods: socio-demographic patient information form, the McGill pain measurement questionnaire and research tracking form will be used.

For pain the McGill pain measurement, for hematoma single use paper tape, for the TR band usage time will be recorded via a chronometer.

For study group I and II patients, cold ball (ISO BALL) application intervention will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* First time receivers of transradial angiography
* Neurovascular extremities must be healthy,
* Must be conscious,
* For the angiography 5 french arterial sheath hydrophylic catheter must be used
* Patients for the study must be voluntary

Exclusion Criteria:

* Unconscious,
* Patients who have unstable Diabetes mellitus,
* Patients who have chronic pain,
* Patients who have carpel tunnel syndrome,
* Patients who have rheumatoid - arthritis,
* Patients who have upper extremity physical disability
* Patients who have any cancer,
* Patients who have bleeding disorders, for example: haemophilia
* Patients who decline to participate in the study.

Patient criteria for study rejection

* Patients who have current chest pain and whose specialist doctor considers their condition too serious for them to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
pain levels | one day
  pain measurement will be made by McGill Pain Survey Short Form. The survey includes visual analog score. The intensity of pain will measure the area in which the individual mark between 0 (no pain) and 10 (worst pain i felt in my life). The pain level will be asked Three times in approximately three hours for all groups patients after transradial angiography
hematoma | one day
  hematoma formation condition will be recorded by single use paper tape measurement for all groups patients. It will be measured three times in approximately three hours after transradial angiography.

SECONDARY OUTCOMES:
Time of Terumo band usage | one day
  time of Terumo band usage will be recorded by chronometer after transradial angiography for all groups patients. Because we want to measure terumo band usage time differences among groups.

CONTACTS AND LOCATIONS:
Overall Officials: atiye erbas, PhD, Principal Investigator — Duzce University

IPD SHARING:
Plan to Share IPD: No